CLINICAL TRIAL: NCT01770951
Title: A Retrospective, Observational, Non-interventional Trial to Assess Eculizumab Treatment Effect in Patients With Atypical Hemolytic Uremic Syndrome (aHUS)
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C09-001r
Record Dates: First submitted 2012-11-13; First posted 2013-01-18 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Atypical Hemolytic Uremic Syndrome (aHUS)
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
The objective of this retrospective trial is to assess safety and efficacy of eculizumab in aHUS patients treated outside of an Alexion-sponsored controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of any age who have been diagnosed with aHUS.
2. Received at least one dose of eculizumab for the treatment of aHUS between 2007 and 2009 outside of an Alexion sponsored controlled clinical trial.

Exclusion Criteria:

1. Patients who have participated or are currently participating in a controlled clinical trial of eculizumab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients of any age who have been diagnosed with aHUS.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2010-11-30 (Actual)

PRIMARY OUTCOMES:
Overall safety and tolerability of eculizumab based on Adverse Events of Special Interest/Adverse Drug Reactions and Additional Adverse Events. | Through 26 weeks

SECONDARY OUTCOMES:
Assess eculizumab treatment affect based on change in laboratory parameters (platelets, hemoglobin, LDH and parameters associated with renal function and intravascular hemolysis) and reduction of thrombotic microangiopathy (TMA). | Through 26 weeks

CONTACTS AND LOCATIONS:
Locations (23):
- United States (12):
  - Dunwoody, Georgia
  - Chicago, Illinois
  - Portland, Maine
  - Boston, Massachusetts
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Corpus Christi, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Spokane, Washington
  - Appleton, Wisconsin
- Austria (2):
  - Graz
  - Innsbruck
- Montreal, Quebec, Canada
- France (3):
  - Caen
  - Le Kremlin-Bicêtre
  - Paris
- Germany (2):
  - Berlin
  - Heidelberg
- Amsterdam, Netherlands
- Barcelona, Spain
- Bern, Switzerland